CLINICAL TRIAL: NCT05626530
Title: A Pilot Trial of the Tolerability and Clinical Effectiveness of Letermovir When Used for Secondary Prophylaxis to Prevent Recurrent Cytomegalovirus Disease in Solid Organ Transplant Recipients
Brief Title: Letermovir for Secondary Prophylaxis in Solid Organ Transplant Recipients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00003219
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cytomegalovirus Infections; Infection in Solid Organ Transplant Recipients; Neutropenia; Antiviral Toxicity
Keywords: Cytomegalovirus infection; Letermovir; Secondary prophylaxis; T cell immunity; neutropenia
MeSH Terms: conditions — Cytomegalovirus Infections; Neutropenia | interventions — letermovir; Bulk Drugs

STUDY DESIGN:
Intervention Model Description: Open label trial of letermovir given to eligible patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Other): This is an open label single arm study
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Open label 480 mg given daily for 60 days
  Other Names: Active drug

SUMMARY:
This is a research study to test the tolerability and clinical effectiveness of the study drug, Letermovir (LET), when used as secondary prophylaxis following treatment of Cytomegalovirus (CMV) infection and disease in a solid organ transplant recipient.

This study is an open label trial in which Letermovir will be prescribed to prevent the recurrence of CMV infection and disease in a solid organ transplant recipient following treatment of CMV infection or disease.

DETAILED DESCRIPTION:
This study will enroll solid organ transplant recipients who develop cytomegalovirus infection and disease who have been treated. At the time of finishing treatment, if the clinician feels that secondary prophylaxis is indicated, they will be enrolled to receive Letermovir 480 mg orally once a day for 60 days. CMV specific T cell assays will be obtained at the initiation of secondary prophylaxis and at the discontinuation of secondary prophylaxis. Patients will be followed for 4 months following discontinuation of secondary prophylaxis to see if they relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (> 18 years old) solid organ transplant recipients (heart, kidney or liver patients) recovering from treated CMV disease in whom the clinician deems that the patient need secondary prophylaxis and in whom written informed consent is obtained.
2. Patient able to participate with follow up for 6 months
3. Not enrolled in competing clinical trials

Exclusion Criteria:

1. Patients with creatinine clearance less than 10 ml per min at time of enrollment
2. Hypersensitivity to letermovir or has a CMV isolate which is known to be resistant to letermovir based on prior testing
3. On CVVH or renal dialysis at the time of enrollment
4. Has Child Pugh Class C severe hepatic insufficiency at screening.
5. Has both moderate hepatic insufficiency AND moderate to severe renal insufficiency at screening.

   Note: Moderate hepatic insufficiency is defined as Child Pugh Class B (Appendix 8); moderate to severe renal insufficiency is defined as CrCl <50 mL/min, as calculated by the Cockcroft-Gault equation.
6. Has a history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ; or is under evaluation for other active or suspected malignancy.
7. Is pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through at least 90 days following cessation of study therapy.
8. Is expecting to donate eggs or sperm starting from the time of consent through at least 90 days following cessation of study therapy.
9. Has a history or current evidence of any condition, therapy, lab abnormality, or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or put the participant at undue risk, as judged by the investigator, such that it is not in the best interest of the participant to participate in this study.
10. Is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within the 6 months) of drug or alcohol abuse or dependence.

    Note: Participants with a history of marijuana use which is not deemed excessive by an investigator or does not interfere with the participant's daily function may participate in the study.
11. Is currently participating or has participated in a study with an unapproved investigational compound or device within 28 days, or 5× half-life of the investigational compound (excluding monoclonal antibodies), whichever is longer, of initial dosing on this study. Participants previously treated with an investigational monoclonal antibody will be eligible to participate after a 150-day washout period.
12. Has previously participated or is currently participating in any study involving administration of a CMV vaccine or another CMV investigational agent that is not approved or is planning to participate in a study of a CMV vaccine or another unapproved CMV investigational agent during the course of this study.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Rate of Relapse after prophylaxis | 6 months after starting intervention
  Proportion of patients with relapsing CMV disease up to 6 months after starting drug

SECONDARY OUTCOMES:
Opportunistic infection | 6 months after starting
  Rate of opportunistic infections or other infectious outcomes in the letermovir arm.
Adverse events associated with taking letermovir | 6 months after starting
  Tolerability and compliance of patients taking letermovir in terms of adverse events
Neutropenia | 6 months after starting intervention
  Duration and nadir of neutropenia in the letermovir group
Rejection | 6 months
  Rate of rejection at 6 months after starting secondary prophylaxis in the letermovir arm.
T cell function | 6 months after starting intervention
  Proportion of patients who have demonstrated CMV specific T cell immunity at start of letermovir secondary prophylaxis will be compared to the proportion who have CMV specific T cell function at the discontinuation of prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Chow, MD, MS, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center-Division of Geographic Medicine and Infectious Diseases, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No